CLINICAL TRIAL: NCT00002652
Title: A PHASE II PILOT STUDY OF SURAMIN IN PREVIOUSLY TREATED PATIENTS WITH MULTIPLE MYELOMA AND PATIENTS WITH CASTLEMAN'S DISEASE
Brief Title: Suramin in Treating Patients With Refractory or Relapsed Multiple Myeloma or Castleman's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000064185; UARK-94016; NCI-T94-0176O
Record Dates: First submitted 1999-11-01; First posted 2004-03-01 (Estimated); Last update posted 2013-02-04 (Estimated); Status verified 2002-04

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: refractory multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Suramin

INTERVENTIONS:
Drug: suramin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of suramin in treating patients who have refractory or relapsed multiple myeloma or Castleman's disease.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the tumor response of patients with refractory or relapsed multiple myeloma or Castleman's disease treated with suramin. II. Determine the effects of this regimen on cytokine-mediated symptoms in patients with Castleman's disease. III. Determine the overall and progression-free survival in patients with multiple myeloma or Castelman's disease treated with this regimen. IV. Determine the qualitative, quantitative, and cumulative toxic effects of this regimen in these patients. V. Determine the effect of this regimen on the levels of serum interleukin-6 (IL-6), soluble IL-6 receptor, and soluble gp130 in these patients.

OUTLINE: Patients receive suramin on days 1-5, 8, 11, 15, 19, 22, and 29. During course 1, patients also receive suramin on days 36, 43, 50, 57, 64, 71, and 78. Suramin is administered IV over 2 hours on day 1 of course 1 and over 1 hour on all subsequent infusion days. Patients undergo rest for at least 12 weeks between each course. Patients with responding disease after completion of course 2 may receive additional courses in the absence of unacceptable toxicity. Patients are followed weekly for 1 month, every 2 weeks for 1 month, at 3 months, and then monthly thereafter if indicated.

PROJECTED ACCRUAL: A total of 20-40 patients with multiple myeloma will be accrued for this study within 10-20 months. A total of 20-40 patients with Castleman's disease will be accrued for this study within 2.9-8 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Confirmed diagnosis of active multiple myeloma Refractory (less than a partial response) to or relapsed after standard chemotherapy Myeloma protein present for response evaluation Nonsecretory myeloma eligible if plasmacytosis greater than 30% OR Pathologic diagnosis of Castleman's disease Multicentric or symptomatic disease requiring therapy Measurable or evaluable disease

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Zubrod 0-2 Life expectancy: At least 1 year Hematopoietic: Absolute granulocyte count greater than 1,500/mm3 Platelet count greater than 100,000/mm3 Hepatic: Bilirubin normal SGOT no greater than 2 times upper limit of normal PT and PTT normal No coagulopathy Renal: Creatinine less than 1.5 mg/dL OR Creatinine clearance greater than 70 mL/min Calcium no greater than 12 mg/dL Other: No severe psychiatric disorder that would preclude informed consent No known seizure disorder No peripheral neuropathy or POEMS (polyneuropathy, organomegaly, endocrinopathy, monoclonal gammopathy, and skin changes) syndrome No uncontrolled or brittle diabetes mellitus HIV negative No other active medical illness that would preclude study No other malignancy within the past 5 years except nonmelanomatous skin cancer or stage IA cervical carcinoma Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception during and for 6 months after study

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 4 weeks since prior biologic therapy Chemotherapy: See Disease Characteristics At least 4 weeks since prior chemotherapy (6 weeks since prior mitomycin or nitrosoureas) Endocrine therapy: At least 4 weeks since prior glucocorticoids (e.g., prednisone, dexamethasone) Radiotherapy: At least 4 weeks since prior radiotherapy No prior radiotherapy to more than 20% of bone marrow Surgery: At least 4 weeks since prior surgery Other: Recovered from the toxic effects of prior therapy No other concurrent therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1995-05; Study Completion 2004-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nikhil C. Munshi, MD, Study Chair — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States